CLINICAL TRIAL: NCT04052204
Title: A Phase 1b/2 Study to Evaluate Safety and Clinical Activity of Avelumab in Combination With Bempegaldesleukin(NKTR-214) With or Without Talazoparib or Enzalutamide in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: Avelumab With Bempegaldesleukin With or Without Talazoparib or Enzalutamide in Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study prematurely terminated as the experimental treatments evaluated in study B9991040 may not provide additional clinical benefit over current or future Standard of Care in the different therapeutic indications that this trial was to evaluate.
Sponsor: Pfizer (Industry)
Collaborators: EMD Serono (Industry); Nektar Therapeutics (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B9991040; 2019-001358-24 (EudraCT Number)
Record Dates: First submitted 2019-08-02; First posted 2019-08-09 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck (SCCHN); Metastatic Castration Resistant Prostate Cancer (mCRPC)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — avelumab; bempegaldesleukin; talazoparib; enzalutamide

STUDY DESIGN:
Intervention Model Description: Combination A: Avelumab + Bempegaldesleukin (NKTR-214) for treatment of locally recurrent (not amendable for treatment with curative intent) or metastatic squamous cell carcinoma of the head and neck
  Combination B: Avelumab + Bempegaldesleukin (NKTR-214) + Talazoparib for treatment of metastatic castration-resistant prostate cancer (mCRPC). Phase 2 will enroll participants with DDR defect positive mCRPC.
  Combination C: Avelumab + Bempegaldesleukin (NKTR-214) + Enzalutamide for Treatment of mCRPC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Combination A (Experimental): Avelumab + Bempegaldesleukin (NKTR-214) for treatment of locally recurrent (not amendable for treatment with curative intent) or metastatic squamous cell carcinoma of the head and neck
  Interventions: Drug: avelumab; Drug: Bempegaldesleukin
- Combination B (Experimental): Avelumab + Bempegaldesleukin (NKTR-214) + Talazoparib for treatment of metastatic castration-resistant prostate cancer (mCRPC). Phase 2 will focus on enrolling participants with DDR defect positive mCRPC.
  Interventions: Drug: avelumab; Drug: Bempegaldesleukin; Drug: talazoparib
- Combination C (Experimental): Combination C: Avelumab + Bempegaldesleukin (NKTR-214) + Enzalutamide for Treatment of mCRPC
  Interventions: Drug: avelumab; Drug: Bempegaldesleukin; Drug: enzalutamide

INTERVENTIONS:
Drug: avelumab — Investigational fully human anti-PD-L1 monoclonal antibody
  Other Names: Bavencio; MSB0010718C
Drug: Bempegaldesleukin — Investigational CD122-biased cytokine agonist
  Other Names: NKTR-214
Drug: talazoparib — poly (adenosine diphosphate [ADP] ribose) polymerase (PARP) inhibitor
  Other Names: Talzenna
  Arms: Combination B
Drug: enzalutamide — androgen receptor inhibitor
  Other Names: Xtandi
  Arms: Combination C

SUMMARY:
Evaluation of the combination of avelumab + bempegaldesleukin (NKTR-214 ) in locally advanced squamous cell carcinoma of the head and neck ( metastatic SCCHN) and avelumab + bempegaldesleukin (NKTR-214) + talazoparib or enzalutamide in metastatic castration resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
Phase 1b/ Phase 2 Design

Phase 1b will be the sequential dose-finding study.

Once the Phase 1b component is completed, Phase 2 will be initiated to further evaluate the safety and anti-tumor activity across combinations of therapy.

Combination A will enroll participants with SCCHN.

Combination B and C will enroll participants with mCRPC

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years old.
* Participants with SCCHN or mCRCP.
* Participants must have histological diagnosis of solid tumors and provide tumor tissue.
* Measurable disease by RECIST v1.1 with at least 1 measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
* Adequate bone marrow, renal and liver function
* Highly effective contraceptive use by men with the ability to father a child or women of childbearing potential.
* A WOCBP must have a negative highly sensitive pregnancy test ([urine or serum] as required by local regulations) at C1D1.
* Signed and dated informed consent.

Exclusion Criteria:

* Known prior severe hypersensitivity to investigational products or any component in their formulations, including known severe hypersensitivity reactions to monocolonal antibodies.
* Known history of: immune-mediated colitis, inflammatory bowel disease, pneumonitis, or pulmonary fibrosis.
* Active or prior autoimmune disease that might deteriorate when receiving an immunostimulatory agent.
* Prior organ transplantation including allogenic stem cell transplantation.
* Vaccination within 4 weeks prior to C1D1 and while on trial is prohibited except for administration of inactivated vaccines.
* Known symptomatic brain lesions requiring steroids.
* Known history of testing positive for human immunodeficiency virus (HIV or known acquired immunodeficiency syndrome (AIDS).
* Positive HBV surface antigen or HCV test indicating acute or chronic infection..
* Active infection requiring systemic therapy
* Clinically significant (i.e., active) cardiovascular disease including the following: documented left ventricular ejection fraction (LVEF) <50% by ECHO/MUGA; cerebral vascular accident/stroke or transient ischemic attack; myocardial infarction; unstable angina; congestive heart failure or serious cardiac arrhythmia (uncontrolled, clinically significant) requiring medication.
* Diagnosis of any other malignancy within 2 years prior to C1D1, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or of the cervix and for Combination A only, low-grade (Gleason 6 or below) prostate cancer on surveillance with no plans for treatment intervention (e.g., surgery, radiation, or castration) or adequately treated prostate cancer.
* Current use of immunosuppressive medication at the time of study enrollment.
* Major surgery within 4 weeks prior to study enrollment.
* Conditions that may impair intake or absorption such as inability to swallow capsules or tablets; known malabsorption syndrome; or baseline diarrhea ≤ Grade 1.
* Participation in other studies involving investigational drug(s) within 2 weeks prior to C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- University of Rochester Medical Center, Rochester, New York, United States
- GZA Ziekenhuizen campus Sint-Augustinus, Wilrijk, Antwerpen, Belgium
- Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship, Poland
- Spain (2):
  - Hospital Quirón Barceloma, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991040

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants screened for this study, 1 of the 4 participants was a screen failure, 3 participants were enrolled and received study treatment in Combination A.
Groups:
- Avelumab + Bempegaldesleukin (NKTR-214) (Combination A): NKTR-214 was administered prior to avelumab. NKTR-214 0.006 mg/kg was administered intravenously (IV) over 30 minutes every 2 weeks (Q2W). Avelumab 800 mg as a 1-hour IV infusion was administered after the NKTR-214 Q2W, at the investigational site on an outpatient basis on Day 1 and Day 15 of each 28-day cycle. Within the 2-day window, avelumab and NKTR-214 were administered on the same day. Dose reduction of NKTR-214 to 0.003 mg/kg Q2W was triggered if higher than expected toxicity is observed at the higher dose (risk of excessive toxicity ≥ 0.25).
- Avelumab + NKTR-214+ Talazoparib (Combination B): The dose level for avelumab was fixed at 800 mg Q2W. The starting dose level for NKTR-214 and talazoparib was determined at the completion of the dose finding for Combination A based on available clinical data. The lowest allowed dose for NKTR-214 was 0.003 mg/kg and the lowest allowed dose for talazoparib was 0.5 mg once daily, in which case participants with moderate renal impairment cannot be enrolled. NKTR-214 was administered prior to avelumab. Talazoparib was taken at the clinic after all procedures/assessments completed, before or after the NKTR-214 and avelumab infusions.
  Arm was not tested as company terminated this study on 21 May 2021.
- Avelumab + NKTR- 214 + Enzalutamide (Combination C): The dose level for avelumab was fixed at 800 mg Q2W. The starting dose level for NKTR-214 and enzalutamide was determined at the completion of the dose finding for Combination A based on available clinical data. The approved label dose for enzalutamide was 160 mg once daily (QD) unless unexpected safety issues requiring it lowering according to the Bayesian Logistic Regression Model (BLRM) recommendation. NKTR-214 was administered prior to avelumab. The daily dose of enzalutamide was taken at the clinic after all procedures/assessments completed, and before or after the avelumab and NKTR-214 infusions.
  Arm was not tested as company terminated this study on 21 May 2021.
Period: Overall Study
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A) | Avelumab + NKTR-214+ Talazoparib (Combination B) | Avelumab + NKTR- 214 + Enzalutamide (Combination C)
Started | 3 | 0 (Arm was not tested due to study termination.) | 0 (Arm was not tested due to study termination.)
Completed | 0 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Progressive disease | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 64.00 [56.0 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: DLTs were graded according to NCI- CTCAE version 4.03 and coded using the latest version of Medical Dictionary for Regulatory Activities (MedDRA) preferred term (PT) as event category and MedDRA primary system organ class (SOC) body term as Body System category.
Time Frame: Cycle 1 of the treatment period (28 days)
Population: The DLT-evaluable analysis set included all enrolled participants in Phase 1b who receive at least one dose of the combination treatment and either experience DLT during the first cycle (28 days) of treatment, or complete the DLT observation period for the first cycle of treatment without a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Duration of Response (DR)
Description: DR was defined, for participants with a confirmed Objective Response (OR), as the time from the first documentation of OR to the date of first documentation of progressive disease (PD) or death due to any cause. The documentation of PD was defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. If a subject had not had an event (PD or death), DR was censored at the date of last adequate tumor assessment.
  As there were no objective responses in the study, no participant met the definition of analysis population.
Time Frame: Approximately 8 months (246 days).
Population: All participants treated in combination A who achieved an OR.
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR was defined, for participants with objective response, as the time from the date of first dose of study treatment to the first documentation of objective response (Complete Response or Partial Response) which was subsequently confirmed.
  As there were no objective responses in the study, no participant met the definition of analysis population.
Time Frame: Approximately 8 months (246 days).
Population: All participants treated in combination A who achieved an OR.
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) was defined as the time from the date of first dose of study treatment to the date of the first documentation of PD or death due to any cause, whichever occurred first. PFS data were censored on the date of the last adequate tumor assessment for participants who did not have an event (PD or death), for participants who started new anti-cancer therapy prior to an event, or for participants with an event after two or more missing tumor assessments. Participants who did not have an adequate baseline tumor assessment or who did not have any adequate post-baseline tumor assessments were censored on the date of first dose of study treatment unless death occurred on or before the time of the second planned tumor assessment, in which case the death was considered an event. PFS time was summarized using the Kaplan-Meier method.
Time Frame: Approximately 8 months (246 days).
Population: All participants treated in Combination A.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
months | 1.69752 [0.59913 to 1.69752]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from the date of first dose of study treatment to the date of death due to any cause. Participants last known to be alive were censored at date of last contact.
  OS time was summarized using the Kaplan-Meier method.
Time Frame: Approximately 8 months (246 days).
Population: All participants treated in Combination A.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
months | 2.56293 [0.59913 to NA] — The upper limit of 95% CI can not be estimated due to small number of events.

6. Secondary Outcome: Pharmacokinetic (PK) Parameters - Cmax and Ctrough for Avelumab and NKTR-214
Description: Cmax was defined as the maximum observed plasma concentration at the end of infusion. Ctrough was defined as the predose concentration at the end of dosing interval.
Time Frame: Blood samples were collected on Day 1 and Day 15 in Cycle 1 and Cycle 2 for avelumab. Blood samples were collected on Day 1, Day 3, Day 4 and Day 8 in Cycle 1, Day1 and Day 8 in Cycle 2 for NKTR-214.
Population: The PK parameter analysis set was a subset of the safety analysis set and included participants who had at least one of the PK parameters of interest for avelumab, NKTR-214, IL-2, talazoparib, enzalutamide, or N-desmethyl-enzalutamide.
Measure: Median (95% Confidence Interval); unit: ug/mL
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
ug/mL | NA [NA to NA] — There were no summaries and interpretations of PK results available, because N<=3 in the PK analysis set.

7. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) Results
Description: ADA against avelumab and NKTR-214 in serum samples was determined and reported separately for ADA never-positive, ADA ever-positive participants, baseline ADA positive, treatment-boosted ADA, treatment-induced ADA, transient ADA response, persistent ADA response. For all participants, blood for ADA samples was drawn from the contralateral arm of the avelumab and NKTR-214 infusion.
Time Frame: Day 1 of Cycle 1, 2 and end of treatment (EOT).
Population: The immunogenicity analysis set was a subset of the safety analysis set and included participants who had at least one ADA/nAb sample collected for avelumab, NKTR-214, or IL-2.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
Participants | NA — ADA results were not analyzed for this study due to study termination.

8. Secondary Outcome: Number of Participants With Positive Neutralizing Antibody (nAb) Results
Description: nAb in serum samples was determined and reported separately for nAb never-positive, nAb ever-positive, baseline nAb positive, treatment-induced nAb, transient nAb response, persistent nAb response.
Time Frame: Day 1 of Cycle 1, 2 and EOT
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
Participants | NA — NAb results were not analyzed for this study due to study termination.

9. Secondary Outcome: PD-L1 Expression Level in Baseline and On-treatment Tumor Tissue
Description: PD-L1 expression level in baseline tumor tissue, and in on-treatment tumor tissue was defined as the number of PD-L1 positive cells and/or qualitative assessment of PD-L1 staining on tumor and/or inflammatory cells in regions of interest. PD-L1 expression level in baseline tumor tissue and in on-treatment tumor tissue were under pathological analyses, assisted by image analysis. Participants were classified as positive or negative according to scoring algorithms and cut-offs established from internal or external sources.
Time Frame: On-treatment biopsy is required to be collected on Cycle 1 between Days 9 and 14 for participants in Combination A.
Population: The biomarker analysis set for biomarkers that were only measured at screening was a subset of the safety analysis set and included participants who had at least one baseline biomarker assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
Participants | NA — No biomarker data (PD-L1) were analyzed for this study due to early study termination.

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events(TEAEs), Serious TEAEs, TEAEs Leading to Death and Infusion-Related Reactions (IRRs) During On-treatment Period
Description: Adverse events (AEs) were any untoward medical occurrences in a participant or clinical study participants, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-emergent adverse events (TEAEs) were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as the time from the first dose of study treatment through minimum (30 days + last dose of study treatment). A Serious Adverse Event (SAE) was defined as any untoward medical occurrence that, at any dose: a. Results in death, b. Was life-threatening, c. Required inpatient hospitalization or prolongation of existing hospitalization, d. Resulted in persistent disability/incapacity, e. Was a congenital anomaly/birth defect. Causality to study treatment was determined by the investigator.
Time Frame: Approximately 6 months (190 days)
Population: The safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
Participants
  Participants with all-causality TEAEs | 3
  Participants with grade ≥ 3 all-causality TEAEs | 2
  Participants with treatment-related TEAEs | 3
  Participants with grade ≥ 3 treatment-related TEAEs | 1
  Participants with serious all-causality TEAEs | 1
  Participants with serious treatment-related TEAEs | 1
  Participants with all-causality TEAEs leading to death | 1
  Participants with treatment-related TEAEs leading to death | 1
  Participants with IRRs | 0

11. Secondary Outcome: Number of Participants With Laboratory Abnormalities With NCI-CTCAE Grade >= 3 - Safety Analysis Set
Description: Liver Function Tests of alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin (TBILI) were used to assess possible drug induced liver toxicity. The number of participants with at least one of the following laboratory results were summarized below: 1. (ALT ≥3 × ULN or AST ≥3 × ULN) post-baseline. 2. TBILI ≥2 × ULN post-baseline. 3. (ALP ≤2 × ULN or missing) post-baseline.
Time Frame: Day 1, Day 15 of each treatment cycle
Population: The safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Approximately 8 months (246 days) . For all causality death cases, all death cases were reported regardless if the cases happened during on-treatment period or not. In total, 2 death cases were reported. Only 1 of the 2 death cases was caused by an adverse event , the other participant died due to disease progression. Thus only 1 serious adverse event was reported. All other reported adverse events are treatment-emergent adverse events.
Arm/Group | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A)
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A) (N=3)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab + Bempegaldesleukin (NKTR-214) (Combination A) (N=3)
Asthenia (General disorders) | 1 (4)
Fatigue (General disorders) | 1 (7)
General physical health deterioration (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (6)
Hypotension (Vascular disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Phase 1b part of Combination A was conducted but not completed as company terminated this study on 21 May 2021. Termination was not due to a regulatory request or new emerging safety signals. Test for Combination B, Combination C and Phase 2 expansion for Combination A planned in the protocol were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT04052204/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT04052204/SAP_001.pdf